CLINICAL TRIAL: NCT03692286
Title: Assessment of Postoperative Pain After Using Silver Nanoparticles With and Without Calcium Hydroxide as an Intracanal Medication in Patients With Necrotic Pulp: (A Randomized Clinical Trial)
Brief Title: Assessment of Postoperative Pain After Using Various Intracanal Medication in Patients With Necrotic Pulp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermine Elsayed Abdelsalam Hassan, Assistant Lecturer of Endodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO18
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Calcium Hydroxide; colloidal silver

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AgNP/Ca(OH) (Active Comparator): Patients receiving combined Silver nanoparticle/Calcium hydroxide administered as intracanal medication at the first visit after cleaning and shaping
  Interventions: Combination Product: Silver nanoparticle/Calcium hydroxide
- AgNP (Active Comparator): Patients receiving silver nanoparticles in gel form administered as intracanal medication at the first visit after cleaning and shaping
  Interventions: Drug: Silver Nanoparticles in gel form
- Ca(OH) (Active Comparator): Patients receiving calcium hydroxide intracanal medication at the first visit after cleaning and shaping
  Interventions: Drug: Calcium Hydroxide Intracanal medication

INTERVENTIONS:
Combination Product: Silver nanoparticle/Calcium hydroxide — Intracanal Medication composed of combined silver nanoparticles with calcium hydroxide
  Arms: AgNP/Ca(OH)
Drug: Silver Nanoparticles in gel form — Intracanal medication composed of silver nanoparticles in gel form
  Arms: AgNP
Drug: Calcium Hydroxide Intracanal medication — Calcium hydroxide intracanal medication
  Arms: Ca(OH)

SUMMARY:
To assess the Postoperative Pain after using Silver Nanoparticles with and without Calcium Hydroxide as an Intracanal Medication in Patients with necrotic pulp (RCT)

DETAILED DESCRIPTION:
When the treatment itself appears to initiate the onset of pain and/or swelling, the result can be very distressing to both the patient and the operator. Patients might even consider postoperative pain and flare-up as a benchmark against which the clinician's skills are measured. Prevalence of postoperative pain or flare-up is, therefore, one of the influencing factors when making a clinical decision. Better management of postoperative pain increases the patients' confidence in dentist's skills and gives positive attitude toward dental profession. In cases with necrotic pulp, the incidence of pain becomes higher, hence testing which intracanal medication is more effective in decreasing the bacteria present within the root canal and subsequently pain is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are free from any physical or mental handicapping condition with no underlying systemic disease.
* Non-pregnant females
* Asymptomatic necrotic mandibular single rooted teeth.
* Normal occlusal contact with the opposing teeth.
* Patients accepting to participate in the study.

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If analgesics or antibiotics have been administrated by the patient during the past 12 hours preoperatively might alter their pain perception
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation Teeth that shows:
* Association with acute periapical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* No restorability: Hopeless tooth.
* Vital teeth
* Immature teeth
* Radiographic evidence of external or internal root resorption.
* Any criterion, not mentioned in the inclusion criteria

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-09-18 (Actual)

PRIMARY OUTCOMES:
Change in post-operative pain | Intra-appointment and post obturation at 4, 24, 48, 72, 96 hours
  Numerical (0-10)

SECONDARY OUTCOMES:
Intracanal Bacterial count reduction | 1 week
  Quantification of Colony forming units per milliliter of agar medium (CFU/mL)
Number of analgesic tablets taken by the patient after endodontic treatment | Within 4 days after the first session and after 1 week from first treatment session
  Number

CONTACTS AND LOCATIONS:
Overall Officials: Nermine Hassan, Msc, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be made available
Supporting Information: Study Protocol, ICF
Time Frame: It will be available after finishing the study
Access Criteria: It will be uploaded on a folder on google drive to be accessed through this link
URL: https://drive.google.com/open?id=1rZXDbSgsneWDO4xGz8KGkklEHHw2YYIX

REFERENCES:
- [Background] Singh RD, Khatter R, Bal RK, Bal CS. Intracanal medications versus placebo in reducing postoperative endodontic pain--a double-blind randomized clinical trial. Braz Dent J. 2013;24(1):25-9. doi: 10.1590/0103-6440201302039. PMID 23657409